CLINICAL TRIAL: NCT02126514
Title: A Phase I, Open-Label, Single-Center Study to Assess the Absorption, Metabolism, and Excretion After Oral Administration of [14C]-AZD3293 to Healthy Male Subjects
Brief Title: A Phase I, Open-Label, Single-Center Study to Assess the Absorption, Metabolism, and Excretion of [14C]-AZD3293
Acronym: AZD3293hADME
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: D5010C00007; AZD3293 hADME (Other: AstraZeneca)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers; Mass Balance Study
Keywords: Beta secretase inhibitor; Alzheimer disease
MeSH Terms: conditions — Alzheimer Disease | interventions — lanabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD3293 (Experimental): 7 subjects will receive AZD3293
  Interventions: Drug: AZD3293

INTERVENTIONS:
Drug: AZD3293 — 7 subjects will receive AZD3293

SUMMARY:
This study will be an open-label, non-randomized, absorption, metabolism, and excretion study to evaluate the mass balance, metabolite profiles, and rates and routes of elimination of [14C]-AZD3293 and derived metabolites following administration as a single 100-mg (containing approximately 150 µCi) oral dose (as an oral solution)

DETAILED DESCRIPTION:
This study will be an open-label, non-randomized,absorption, metabolism, and excretion study to evaluate the mass balance, metabolite profiles, and rates and routes of elimination of [14C]-AZD3293 and derived metabolites following administration as a single 100-mg (containing approximately 150 µCi) oral dose (as an oral solution) following at least an 8-hour fast from food (not including water). Seven healthy male subjects will be enrolled in the study at a single study site to complete a minimum of 6 subjects. The study will consist of 2 visits.

ELIGIBILITY:
Inclusion Criteria: Healthy male subjects between 18 and 55 years of age, inclusive, at the time of consent with suitable veins for cannulation or repeated venipuncture; 2) Body weight between 50 to 100 kg, inclusive; 3) Within BMI range 19 to 30 kg/m2, inclusive; 4) In good health, as determined by no clinically significant findings from medical history, physical examination with neurological examination, 12-lead ECG, and vital signs as judged by the Investigator;

-

Exclusion Criteria:

Participation in any prior study of AZD3293 or previous enrollment in the present study; 2) Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, interfere with absorption, distribution, metabolism or excretion of drugs, or influence the results or the subject's ability to participate in the study; 3) History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator;

-

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
PK parameters measured by assessment of AUC over time and Maximum observed concentration (Cmax) | Up to Day 25
  Maximum observed concentration (Cmax) parameters will be calculated, for AZD3293, its metabolite; and [14C]-AZD3293-derived total radioactivity.

SECONDARY OUTCOMES:
Safety assessments including vital sign measurements, ECGs, physical examinations, clinical laboratory evaluations, and a record of adverse events (AEs). | Up to Day 25
  Safety assessments including vital sign measurements, ECGs, physical examinations, clinical laboratory evaluations, and a record of adverse events (AEs), will be performed before and following investigational product administration.
The Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to day 25
  The Columbia-Suicide Severity Rating Scale (C-SSRS) will be used to assess the psychiatric health of subjects.
Time to maximum observed concentration (tmax) | Up to day 25
  Time to maximum observed concentration (tmax) will be calculated for AZD3293 and its metabolite; and [14C]-AZD3293-derived total radioactivity.
Area under the concentration-time curve | Up to day 25
  Area under the concentration-time curve from Hour 0 to the last measurable concentration (AUC0-t), will be calculated for AZD3293 and its metabolite ; and [14C]-AZD3293-derived total radioactivity concentrations.
Area under the concentration-time curve extrapolated to infinity (AUC0-∞) | Up to day 25
  Area under the concentration-time curve extrapolated to infinity (AUC0-∞), apparent terminal elimination rate constant (λZ), will be calculated for AZD3293 and its metabolite ; and [14C]-AZD3293-derived total radioactivity.
Apparent terminal elimination half-life (t1/2) | Up to day 25
  Apparent terminal elimination half-life (t1/2), will be calculated for AZD3293 and its metabolite; and [14C]-AZD3293-derived total radioactivity.
Apparent oral clearance (CL/F) | Up to day 25
  Apparent oral clearance (CL/F) (AZD3293 only), will be calculated for AZD3293 concentrations.
Apparent volume of distribution (Vz/F) | Up to day 25
  Apparent volume of distribution (Vz/F) (AZD3293 only) will be calculated for AZD3293 concentrations.
Ratios for AUC0- | Up to day 25
  Ratios for AUC0- including the ratio of total radioactivity in whole blood/plasma; and the ratio of AZD3293 in plasma and total radioactivity in plasma, will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Irene Mirkin, MD, Principal Investigator — Covance
Locations (1):
- Research Site, Madison, Wisconsin, United States